CLINICAL TRIAL: NCT04618172
Title: Effects of Exercise on the Symptoms of Premenstrual Syndrome and Dysmenorrhoea and Blood Flow of Genital Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kovács Zoltán (Other)
Responsible Party: Sponsor-Investigator, Kovács Zoltán, Principal Investigator, University of Pecs
Organization: University of Pecs (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRKZ01
Record Dates: First submitted 2020-10-19; First posted 2020-11-05 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Premenstrual Syndrome; Dysmenorrhoea
MeSH Terms: conditions — Premenstrual Syndrome; Dysmenorrhea | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Effects of exercise on the symptoms of premenstrual syndrome and dysmenorrhoea and blood flow of genital tract. Different self-reported questionnaires and vaginal ultrasound flowmetry are used in the prospective observational study. The study has interventional and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercising group (Experimental): This group practises 30 minute long exercises twice a week besides filling out the questionnaires.
  Interventions: Other: Exercise
- Control group (No Intervention): This group fills out the questionnaires without practising 30 minute long exercises twice a week.

INTERVENTIONS:
Other: Exercise — 30 minute long exercises twice a week
  Arms: Exercising group

SUMMARY:
Effects of exercise on the symptoms of premenstrual syndrome and dysmenorrhoea and blood flow of genital tract. Different self-reported questionnaires and vaginal ultrasound flowmetry are used in the prospective observational trial. The study has interventional and control groups. There are changes in premenstrual syndrome complaints and dysmenorrhoea complaints during the study period.The deegre of menstrual pain and self-awareness improve during the period of study. The ultrasound examination shows changes in genital blood flow after exercise.

DETAILED DESCRIPTION:
Subject of the study:

Examination of premenstrual syndrome and dysmenorrhoea treatment results with Aviva exercise intervention.

Method of the study:

Prospective observational trial with the participation of volunteers.

Questionnaires:

1. PRISM calendar: Prospective Record of the Impact and Severity of Menstrual Symptoms (Reid, 1995). The participants have to fill out this every day,
2. The Body Awareness Questionnaire Shields, S. A., Mallory, M.E., & Simon, A. (1989). The Body Awareness Questionnaire: Reliability and validity. Journal of Personality Assessment, 53(4), 802-815
3. Examination to measure the intensity of menstrual pain: Numeric Rating Scale
4. Heart rate monitoring and documentation before and after the exercises; completion of the Borg Scale of Perceived Exertion to measure exercise intensity;
5. Questionnaire of life style
6. Beck depression questionnaire

Ultrasound examination:

Doing the Aviva exercises, ultrasound measurements are performed in Robert Hospital (Budapest) on the patients participating in the study. The first measurement is performed for each person before starting the exercises. When the first subject has finished the exercise, a control ultrasound measurement will be carried out.

In the control group there is also twice ultrasound examination for the individuals.

Measured parameters: PI (pulsatility index) of uterine artery transvaginal ultrasound measurement followed by statistical evaluation of the results.

ELIGIBILITY:
Inclusion Criteria:

* BMI 17-35
* regular menstrual cycles (cycles of 21-35 days)
* no endocrinological disease
* no endometriosis
* no experience in Aviva aerob exercises
* symptoms of premenstrual syndrome
* symptoms of dysmenorrhoea
* Score below 40 from Beck depression questionnaire

Exclusion Criteria:

* pregnancy
* pelvic inflamatory disease (PID), secondary dysmenorrhoea
* gynecological operation
* failure to complete the questionnaire (3 consecutive days and 5 days interrupted)
* dissatisfaction with the continuation of the research
* the incidence of adverse life events in the last 3 months
* use of medication (e.g. oral birth control pill,painkiller,antipsychotic tablets)
* participation in other sports programs
* congenital uterine anomalies
* any chronic disease (e.g. neurological, psychological disorders, endocrinological diseases)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change of premenstrual syndrome complaints | Change of from baseline premenstrual syndrome complaints at next cycle
  Rate of variation of premenstrual syndrome complaints of the participants presented in PRISM (Prospective Record of the Impact and Severity of Menstrual Symptoms) questionnaire
Change of dysmenorrhoea complaints | Change of from baseline dysmenorrhoea complaints at next cycle
  Rate of variation of dysmenorrhoea complaints of the participants presented in Numeric Rating Scale
Change in the genital blood flow | Change of from baseline art.uterina ultrasound flowmetry results after aerobic exercises and 30 minute long waiting time for control individuals
  PI values of ultrasound flowmetry of uterine arteries presented in charts

SECONDARY OUTCOMES:
Change of body-mind awareness | Change of from baseline body-mind awareness results at the end of the first and second cycle
  Change of body-mind awareness using The Body Awareness Questionnaire
Adherence | up to 2 menstrual cycle
  Measurement of adherence: frequency of visiting exercising group

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Szőke Dr, PhD, Study Chair — University of Pecs
Locations (1):
- Róbert Kórház, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kovacs Z, Hegyi G, Szoke H. The Effect of Exercise on Pulsatility Index of Uterine Arteries and Pain in Primary Dysmenorrhea. J Clin Med. 2023 Nov 10;12(22):7021. doi: 10.3390/jcm12227021. PMID 38002635